CLINICAL TRIAL: NCT00374608
Title: A Single Center, Prospective, Pilot Study Examining the Evaluation of Exercise Capacity in Chronically RV Paced Children and Young Adults
Brief Title: Exercise in Chronically Paced Children
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Patricio A. Frias, MD, Associate Professor, Pediatrics, Emory University
Other Study IDs: 291-2006
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Congenital Diseases; Complete Heart Block; Pacemaker
Keywords: pediatric; congenital complete heart block; dual chamber pacemaker
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Congenital heart block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the exercise capacity of patients with complete heart block who are chronically being paced from the right ventricle. Also, we hope to correlate the level of uncoordinated contraction with the patients exercise capacity. We will enroll patients with complete heart block as diagnosed by standard electrocardiographic means and now have a permanent pacemaker. All patients we approach for this study will receive an echocardiogram to assess their heart function. As part of the echocardiogram, they will also receive a Tissue Synchronization Imaging (TSI) evaluation to assess the level of uncoordinated contraction they have. The patients will then be subjected to a cardiac exercise stress test which will involve them running on a treadmill until they cannot continue while data is collected regarding their heart's response to exercise. All portions of the study are noninvasive, which means they work from probes and monitors outside the body.

DETAILED DESCRIPTION:
In third degree, or complete atrioventricular (AV) block, atrial electrical impulses fail to conduct to the ventricles. Congenital complete AV block (CCAVB) has an incidence of 1 in 15,000 to 1 in 25,000 live births and has a strong association with maternal antibodies. Patients with isolated CCAVB range from completely asymptomatic to experiencing syncope, exercise intolerance or congestive heart failure. A portion of the symptoms attributable to CCAVB are secondary to the inability to increase heart rate, and hence cardiac output, in response to varying physiologic demands. For symptomatic patients, the mainstay of therapy has been cardiac pacing. Dual chamber pacing, with atrial sensing and ventricular pacing, allows for restoration of physiologic heart rates and response to exercise or increased metabolic demands. Resumption of AV synchrony allows for more efficient ventricular filling. Overall, pacing in patients with CCAVB would be expected to result in improved cardiac function and exercise tolerance.

The traditional ventricular site for pacing in patients with CCAVB has been the right ventricular apex (RVA). This results in interventricular dyssynchrony as pacing first stimulates the right ventricle, rather than the typical midline ventricular activation pattern seen in patients with intact AV node conduction. Mounting evidence shows that long term RV pacing results in morphologic changes to the LV with resultant compromised performance. Further studies have shown that chronic RV pacing diminishes exercise capacity in patients with heart failure as well as asymptomatic adults. There have been studies, by our group in particular, that have documented ventricular changes in the paced pediatric patient. No published study has examined the possible deleterious effects of RV pacing on exercise capacity in children. We, therefore, propose to do a detailed evaluation of exercise performance, as measured by exercise duration, maximal heart rate, oxygen uptake and ventilatory response, in asymptomatic chronically RV paced children and young adults.

Specific Aim 1: To describe the effects of dyssynchronous ventricular activation on exercise performance in children requiring long term RV pacing

Hypothesis 1: Long term dyssynchronous electromechanical activation, secondary to right ventricular apical pacing, has deleterious effects on the exercise capacity of asymptomatic pediatric patients.

Specific Aim 2: To correlate changes in exercise performance with tissue Doppler indices of mechanical dyssynchrony.

Hypothesis 2: Tissue Doppler is a sensitive means of evaluating dyssynchrony in chronically paced patients.

Background and Significance The goal of pacemaker therapy for CCAVB is to restore, as closely as can be approximated, physiologic rates and activation. Standard dual chamber pacing allows for sinus node participation in cardiac conduction. As a result, a more physiologic chronotropic response to exercise and AV conduction could be achieved. Indeed, prior studies concluded that dual chambered pacing resulted in increased exercise performance and improved perception of general well being as compared to ventricular demand pacing [1-3]. There is, however, increasing evidence that long term RVA pacing leads to detrimental effects on cardiac function secondary to the non-physiologic ventricular activation sequence. Animal studies have revealed regional left ventricular changes in perfusion, function and innervation in chronically RVA paced subjects as well as asymmetric hypertrophy of the LV wall [4,5]. Examinations of patients with inter/intraventricular dyssynchrony reveal a loss of coordination of ventricular contraction and relaxation. When the RV is the initial site of activation, portions of the LV are prematurely activated resulting in early segmental contraction at a low pressure with dissipation of energy and no resultant ejection, while the areas that activate later do so at higher stress and effect a paradoxical stretch on earlier contracted areas [6]. These factors lead to decreased efficiency and diminished systolic function. Ventricular dyssynchrony impairs LV pressure generation, diastolic filling and stroke volume, as well as, increasing wall stress [7]. Tissue Doppler echocardiography has recently proven to be a valuable tool in assessing and verifying regional wall motion abnormalities and aberrant LV activation by its ability to determine peak systolic velocity of different myocardial regions, degree of myocardial deformation and distinguish between active systolic contraction and passive displacement [8,6].

Recognizing the less-than-optimal long term functional and hemodynamic effects of RVA pacing, prior investigators have attempted to utilize alternative RV pacing sites with variable success in improving LV function [9,10]. Most evidence, however, indicates that dyssynchrony results in maladaptive ventricular remodeling compromised function and decreased exercise capacity [11,12]. Evaluation of patients with dilated cardiomyopathy and conduction delay has yielded ample evidence of the deleterious effects of dysscynchronous ventricular activation. Conversely, the positive response to the restoration of ventricular synchrony via bi-ventricular pacing has further highlighted the negative effects of ventricular dyysynchrony. In this subset of patients, acute biventricular pacing, as compared to RV pacing, demonstrated increases in systolic function and ejection fraction, along with decreased mitral insufficiency and LV volumes [13]. Resynchronization positively influences reverse remodeling with significant reductions in LV end systolic and LV end diastolic volumes and left atrial size - changes that appear permanent [7]. Resynchronization has also been implicated in improved exercise capability, peak oxygen uptake and improved quality of life measures [14].

With established evidence of maladaptive changes to cardiac morphology and function, plus emerging evidence of adversely effected exercise capacity in adults with chronic RVA pacing, it is necessary to investigate the possible aberrancy in exercise capacity in the RVA paced pediatric population.

Patient Population

Patients between 10 and 21 years of age seen at Children's Healthcare of Atlanta and Sibley Heart Center satisfying the following criteria:

* Structurally normal heart
* Congenital complete heart block
* Dual chamber, right ventricular apex paced
* Normal function via traditional transthoracic echocardiography
* Absence of preexisting condition that precludes patient from exercise All participating subjects and their parents (if applicable) will be required to sign an informed consent prior to any study procedure. Patients with repaired or palliated congenital heart disease will be excluded from the study. We anticipate enrolling 30 patients for this study.

Research Design and Methods

Design:

The proposed study will be a single center, prospective, pilot examination of exercise capacity in pediatric patients requiring right ventricular apical pacing. We will assess the effects of chronic ventricular dyssynchrony on exercise duration, oxygen uptake and ventilatory response to exercise. All subjects will be extracted from active patients of the Children's Healthcare of Atlanta/ Sibley Heart Center pacemaker clinic, being followed for CCAVB and dual chamber RVA pacing. All participants will be required to sign an informed consent prior to a procedures. Patients with palliated or corrected congenital heart disease will be excluded.

Procedures:

1. Echocardiographic Assessment: all participants will receive a standard 2-dimensional M-mode and Doppler evaluation. We will assess cardiac function using left ventricular shortening fraction and ejection fractions. Tissue Doppler imaging will be utilized to evaluate ventricular synchrony.
2. Exercise Testing: Using a modified Bruce treadmill protocol, with staged increases in belt speed and incline, the subject's duration of exercise, work, oxygen uptake, maximal heart rate, blood pressure and ventilatory responses will be measured. The procedure will take place at the exercise laboratory at Children's Healthcare of Atlanta at Egleston, utilizing the customary staff. There will be physician attendance for all procedures. Analysis of the exercise results will be conducted by an attending pediatric cardiologist.
3. Clinical Assessment: Clinical evaluation will be performed during routine pacemaker clinic visit, during treadmill exercise testing and at subsequent routine pacemaker clinic visits. The information gained from this study will not be used for individual care.

Study Regimens After eligibility is established and baseline assessment completed, consenting patients will undergo exercise treadmill testing. Using established CHOA protocols, max heart rate, oxygen uptake, blood pressure and ventilatory changes will be measured during the test. Subjects will then return to their usual and customary cardiac follow up schedule.

MANAGEMENT OF ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS

1. Monitoring of Adverse Events (AEs) and Serious Adverse Events (SAEs) is an important aspect of data collection in this study. Families will be questioned about possible AEs follow up survey and asked to notify clinical staff of any AE, illness, medical procedure or hospitalization. The duration after the completion of all study procedures for which AE's will be recorded will be one month. One month will be a sufficient time to capture all possible AE's given that most potential AE's would occur in the immediate testing period. An adverse event case report form (CRF) will be created to capture any medical symptoms experienced since the exercise test to solicit unexpected AEs. For any adverse experience reported during the study, the nature, duration, intensity and any remedial action will be recorded. Serious AEs (life-threatening, requiring hospitalization) will be reported to the IRB within 48 hours of notification. The Research Coordinator in conjunction with the Principal Investigator will collect the adverse experiences from the medical record/subject. The Principal Investigator will determine the seriousness of each adverse event.

Statistical Considerations We anticipate analyzing the obtained data utilizing analysis of covariance (ANCOVA). The independent variable will be the group assignment (healthy vs paced patients) and the co-variable being added to the model is age.

Ethics and Patient Safety This study will be conducted in accordance with the ethical principals that have their base in the Declaration of Helsinki and will be conducted with Good Clinical Practice (GCP) and applicable regulatory requirements. This study will be conducted in compliance with the protocol. The protocol, any amendments and the subject informed consent will receive Institutional Review Board (IRB) approval prior to initiation. During the conduct of the study, all adverse events will be reported to the IRB during the renewal period however, adverse events classified as serious (SAEs) will be reported within 24 hour of knowing of the occurrence to the IRB.

Freely given written informed consent including patient authorization per HIPAA guidelines will be obtained from every subject, parent or legal guardian prior to the initiation of any study procedures. A copy of all consent documents will be provided to the parent or legal guardian. The rights, safety and well-being of the trial subjects are the most important considerations and will prevail over interests of science and society.

ELIGIBILITY:
Inclusion Criteria:

* between 10 and 21 years of age
* structurally normal heart
* congenital complete heart block
* dual chamber pacemaker, right ventricular apex paced
* normal function via traditional transthoracic echocardiography

Exclusion Criteria:

* preexisting condition that precludes patient from exercise
* no informed consent

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pt who have congenital complete heart block with no other preexisting condition that precludes the patient from exercise
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio A Frias, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Ijiri H, Komori S, Kohno I, Sano S, Yin D, Takusagawa M, Iida T, Yamamoto K, Osada M, Sawanobori T, Ishihara T, Umetani K, Tamura K. Improvement of exercise tolerance by single lead VDD pacemaker: evaluation using cardiopulmonary exercise test. Pacing Clin Electrophysiol. 2000 Sep;23(9):1336-42. doi: 10.1111/j.1540-8159.2000.tb00960.x. PMID 11025888
- [Background] Sulke N, Dritsas A, Bostock J, Wells A, Morris R, Sowton E. "Subclinical" pacemaker syndrome: a randomised study of symptom free patients with ventricular demand (VVI) pacemakers upgraded to dual chamber devices. Br Heart J. 1992 Jan;67(1):57-64. doi: 10.1136/hrt.67.1.57. PMID 1739528
- [Background] Lee MA, Dae MW, Langberg JJ, Griffin JC, Chin MC, Finkbeiner WE, O'Connell JW, Botvinick E, Scheinman MM, Rosenqvist M. Effects of long-term right ventricular apical pacing on left ventricular perfusion, innervation, function and histology. J Am Coll Cardiol. 1994 Jul;24(1):225-32. doi: 10.1016/0735-1097(94)90567-3. PMID 8006270
- [Background] Bax JJ, Ansalone G, Breithardt OA, Derumeaux G, Leclercq C, Schalij MJ, Sogaard P, St John Sutton M, Nihoyannopoulos P. Echocardiographic evaluation of cardiac resynchronization therapy: ready for routine clinical use? A critical appraisal. J Am Coll Cardiol. 2004 Jul 7;44(1):1-9. doi: 10.1016/j.jacc.2004.02.055. PMID 15234396
- [Background] Saxon LA, De Marco T, Schafer J, Chatterjee K, Kumar UN, Foster E; VIGOR Congestive Heart Failure Investigators. Effects of long-term biventricular stimulation for resynchronization on echocardiographic measures of remodeling. Circulation. 2002 Mar 19;105(11):1304-10. doi: 10.1161/hc1102.105730. PMID 11901040
- [Background] Waggoner AD, Bierig SM. Tissue Doppler imaging: a useful echocardiographic method for the cardiac sonographer to assess systolic and diastolic ventricular function. J Am Soc Echocardiogr. 2001 Dec;14(12):1143-52. doi: 10.1067/mje.2001.115391. PMID 11734780
- [Background] Wonisch M, Lercher P, Scherr D, Maier R, Pokan R, Hofmann P, von Duvillard SP. Influence of permanent right ventricular pacing on cardiorespiratory exercise parameters in chronic heart failure patients with implanted cardioverter defibrillators. Chest. 2005 Mar;127(3):787-93. doi: 10.1378/chest.127.3.787. PMID 15764758
- [Background] Thambo JB, Bordachar P, Garrigue S, Lafitte S, Sanders P, Reuter S, Girardot R, Crepin D, Reant P, Roudaut R, Jais P, Haissaguerre M, Clementy J, Jimenez M. Detrimental ventricular remodeling in patients with congenital complete heart block and chronic right ventricular apical pacing. Circulation. 2004 Dec 21;110(25):3766-72. doi: 10.1161/01.CIR.0000150336.86033.8D. Epub 2004 Dec 6. PMID 15583083
- [Background] Yu CM, Lin H, Fung WH, Zhang Q, Kong SL, Sanderson JE. Comparison of acute changes in left ventricular volume, systolic and diastolic functions, and intraventricular synchronicity after biventricular and right ventricular pacing for heart failure. Am Heart J. 2003 May;145(5):E18. doi: 10.1016/S0002-8703(03)00071-1. PMID 12766742
- [Background] Cazeau S, Leclercq C, Lavergne T, Walker S, Varma C, Linde C, Garrigue S, Kappenberger L, Haywood GA, Santini M, Bailleul C, Daubert JC; Multisite Stimulation in Cardiomyopathies (MUSTIC) Study Investigators. Effects of multisite biventricular pacing in patients with heart failure and intraventricular conduction delay. N Engl J Med. 2001 Mar 22;344(12):873-80. doi: 10.1056/NEJM200103223441202. PMID 11259720